CLINICAL TRIAL: NCT03181399
Title: Dietary Treatment of Glucose Transporter Type 1 Deficiency (G1D)
Brief Title: Diet Treatment Glucose Transporter Type 1 Deficiency (G1D)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Juan Pascual, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122016-013; 1R01NS094257-01A1 (NIH)
Record Dates: First submitted 2017-04-25; First posted 2017-06-08 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: GLUT1DS1; Epilepsy; Glut1 Deficiency Syndrome 1, Autosomal Recessive; Glucose Metabolism Disorders; Glucose Transport Defect; Glucose Transporter Type 1 Deficiency Syndrome; Glucose Transporter Protein Type 1 Deficiency Syndrome
MeSH Terms: conditions — Epilepsy; Glucose Metabolism Disorders; Glycogen Storage Disease Id; Glut1 Deficiency Syndrome | interventions — triheptanoin

STUDY DESIGN:
Intervention Model Description: All subjects will receive supplementation at the maximum tolerated dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Triheptanoin (Experimental): This is a single arm study.
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — . Triheptanoin will be taken 4 times per day (approximately every 6 hours: prior to breakfast, lunch and dinner and a mid-afternoon snack) by mouth. It is dosed 4 times per day, divided evenly.
  Other Names: C7

SUMMARY:
Forty-five subjects receiving no dietary therapy with a proven G1D diagnosis will be enrolled. To evaluate the effect of C7 supplementation of a regular diet on a EEG activity in addition to IQ, language, working memory, processing speed, emotional and behavioral functioning, ataxia, and other neuropsychological and neurological performance indices in children and adults genetically diagnosed with G1D receiving a regular diet at enrollment.

DETAILED DESCRIPTION:
This is an open-label, single arm trial of orally-administered C7 in G1D. Subjects will replace a fixed percentage of their daily caloric intake (based on the results of Protocol 1) with C7 for 6 months, undergo full evaluation and discontinuation of treatment at a 6 month visit, and return for an off-treatment follow up visit 3 months after C7 oil discontinuation, for total duration of participation of 9 months. Subjects will undergo treatment initiation on a 24-hour inpatient basis. During that 24-hr inpatient treatment initiation, subjects will have continuous EEG both to monitor for real-time seizure activity (for safety) and to determine EEG changes (secondary outcome) before, during, and after treatment initiation. Subjects will undergo clinical evaluation, comprehensive blood work, ataxia scale rating, EEG, and neuropsychological testing at baseline, 6 months, and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glucose transporter type I deficiency (G1D), confirmed by clinical genotyping at a CLIA-certified laboratory or by PET scan.
* Stable diet on either a modified atkins diet or on no dietary therapy (i.e., no dietary therapy for 1 month).
* Males and females 24 months to 35 years old, inclusive.

Exclusion Criteria:

* Subjects with evidence of independent, unrelated metabolic and/or genetic disease.
* Subjects with a chronic gastrointestinal disorder, such as irritable bowel syndrome, Crohn's disease, or colitis that could increase the subject's risk of developing diarrhea or stomach pain.
* Subjects with a BMI (body mass index) greater than or equal to 30.
* Subjects currently on dietary therapy (i.e., ketogenic diet, medium chain triglyceride supplemented diets, Atkins diet, low glycemic index diet).
* Subjects with no evidence of abnormal EEG (spike wave discharges) in the last 12 months.
* Women who are pregnant or breast-feeding may not participate. Women who plan to become pregnant during the course of the study, or who are unwilling to use birth control to prevent pregnancy (including abstinence) may not participate. Females age 10 and over will be asked to provide a urine sample for a pregnancy test via dipstick. Subjects will be asked to agree to abstinence or another form of birth control for the duration of the study.
* Allergy/sensitivity to C7.
* Previous use of triheptanoin in the past 1 month. Subjects who participate in Protocol 1 of this study are thus eligible.
* Subjects exhibiting signs of dementia, or diagnosed with any degenerative brain disorder (such as Alzheimer's disease) that would confound assessment of cognitive changes, in the opinion of the investigator.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent, or assent for children age 10-17.
* Addition of a new antiseizure drug in the previous 3 months.

Ages: 24 Months to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pascual, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pascual JM, Ronen GM. Glucose Transporter Type I Deficiency (G1D) at 25 (1990-2015): Presumptions, Facts, and the Lives of Persons With This Rare Disease. Pediatr Neurol. 2015 Nov;53(5):379-93. doi: 10.1016/j.pediatrneurol.2015.08.001. Epub 2015 Aug 10. PMID 26341673
- [Background] Hao J, Kelly DI, Su J, Pascual JM. Clinical Aspects of Glucose Transporter Type 1 Deficiency: Information From a Global Registry. JAMA Neurol. 2017 Jun 1;74(6):727-732. doi: 10.1001/jamaneurol.2017.0298. PMID 28437535
- [Background] Pascual JM, Liu P, Mao D, Kelly DI, Hernandez A, Sheng M, Good LB, Ma Q, Marin-Valencia I, Zhang X, Park JY, Hynan LS, Stavinoha P, Roe CR, Lu H. Triheptanoin for glucose transporter type I deficiency (G1D): modulation of human ictogenesis, cerebral metabolic rate, and cognitive indices by a food supplement. JAMA Neurol. 2014 Oct;71(10):1255-65. doi: 10.1001/jamaneurol.2014.1584. PMID 25110966

RESULTS

PARTICIPANT FLOW:
Groups:
- Triheptanoin: This is a single arm study. Patients diagnosed with G1D were enrolled in the study. They received the triheptanoin oil treatment dosed at 45% of the participant's daily caloric intake, divided into 4 doses per day. This intervention was administered for 6 months followed by a 3 month off intervention period.
Period: 6 Months on Treatment
Arm/Group | Triheptanoin
Started | 45
Completed | 29
Not Completed | 16
Not completed — Protocol non-compliance | 7
Not completed — Adverse Event | 4
Not completed — Tried alternative treatment | 2
Not completed — Lost to Follow-up | 2
Not completed — Personal reasons | 1
Period: 3 Months Off-treatment
Arm/Group | Triheptanoin
Started | 29
Completed | 28
Not Completed | 1
Not completed — Parent unable to travel | 1

BASELINE CHARACTERISTICS:
Arm/Group | Triheptanoin
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.53 (5.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychological Score of Sustained Attention
Description: Sustained attention was evaluated using a subtest of Conners' Kiddie Continuous Performance Test Second Edition (K-CPT 2): CPT-Hit Reaction Time Block Change. CPT HRT BC indicates the change in mean response speed as the administration of the test progresses in blocks. A decrease in CPT HRT BC indicates a decrease in reaction time, which means the participant's information processing efficiency increases, and an improvement in sustained attention is noted. The number of participants that showed a decrease in the CPT HRT BC score after 6 months of treatment as compared to baseline is noted here.
Time Frame: Change post 6 months of treatment
Population: Although 29 patients completed the 6-month treatment phase, some patients were unable to perform the test due to cognitive or physical impairment. The analysis population comprises of participants who were present at the time of testing and were able to comprehend and perform the test.
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 16
Participants | 11

2. Primary Outcome: Neuropsychological Score of Sustained Attention
Description: Sustained attention was evaluated using a subtest of Conners' Kiddie Continuous Performance Test Second Edition (K-CPT 2): CPT-Hit Reaction Time Block Change. CPT HRT BC indicates the change in mean response speed as the administration of the test progresses in blocks. A decrease in CPT HRT BC indicates a decrease in reaction time, which means the participant's information processing efficiency increases, and an improvement in sustained attention is noted. The off-treatment period of 3 months was implemented to study whether the impact of treatment persists or goes back to baseline. The number of patients that displayed an increase in CPT HRT BC score (towards baseline) after 3 months off treatment as compared to 6 months on treatment is noted here.
Time Frame: Change after 3 months off treatment
Population: Although 28 patients completed the 3-month treatment phase, some patients were unable to perform the test due to cognitive or physical impairment. The analysis population comprises of participants who were present at the time of testing and were able to comprehend and perform the test.
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 15
Participants | 14

3. Primary Outcome: Neuropsychological Score of Working Memory Index Scale (WMI)
Description: Subjects were administered the Working Memory Index Scale (WMI) from either the Wechsler Primary and Preschool Scale of Intelligence, 4th Edition (WPPSI-IV), Wechsler Intelligence Scale for Children, 5th Edition (WISC-V), or the Wechsler Adult Intelligence Scale, 4th Edition (WAIS-IV) according to the age of subject. An increase WMI score would indicate an improvement in the cognitive ability of identifying, reorganizing and retaining information for a brief period of time. The number of participants that showed an increase in the WMI score after 6 months of treatment is noted here.
Time Frame: Change post 6 months of treatment
Population: Some patients were unable to perform the test due to cognitive, physical impairment or underdeveloped vocabulary skills. The analysis population comprises of participants who were present at the time of testing and were able to comprehend and perform the test.
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 17
Participants | 7

4. Primary Outcome: Neuropsychological Score of Working Memory Index Scale (WMI)
Description: Subjects were administered the Working Memory Index Scale (WMI) from either the Wechsler Primary and Preschool Scale of Intelligence, 4th Edition (WPPSI-IV), Wechsler Intelligence Scale for Children, 5th Edition (WISC-V), or the Wechsler Adult Intelligence Scale, 4th Edition (WAIS-IV) according to the age of subject. An increase WMI score would indicate an improvement in the cognitive ability of identifying, reorganizing and retaining information for a brief period of time. The 3 months off-treatment period was designed to study whether the impact of treatment persists or goes back to baseline. The number of participants that showed a decrease in the WMI score after 3 months off treatment as compared to 6 months on treatment was calculated.
Time Frame: Change after 3 months off-treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 15
Participants | 5

5. Primary Outcome: Neuropsychological Score of Processing Speed Index (PSI)
Description: Subjects were administered the Processing Speed Index Scale (PSI) from either the Wechsler Primary and Preschool Scale of Intelligence, 4th Edition (WPPSI-IV), Wechsler Intelligence Scale for Children, 5th Edition (WISC-V) or the Wechsler Adult Intelligence Scale, 4th Edition (WAIS-IV) according to the age of subject. An increase PSI score would indicate an improvement in the motor-based estimate of the subject's cognitive processing speed. The number of participants that showed an increase in the PSI score after 6 months of treatment as compared to baseline is noted here.
Time Frame: Change post 6 months of treatment
Population: Some patients were cognitively unable to perform or comprehend the test. The analysis population comprises of participants who were present at the time of testing and were able to comprehend and perform the test.
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 15
Participants | 6

6. Primary Outcome: Neuropsychological Score of Processing Speed Index (PSI)
Description: Subjects were administered the Processing Speed Index Scale (PSI) from either the Wechsler Primary and Preschool Scale of Intelligence, 4th Edition (WPPSI-IV), Wechsler Intelligence Scale for Children, 5th Edition (WISC-V) or the Wechsler Adult Intelligence Scale, 4th Edition (WAIS-IV) according to the age of subject. An increase PSI score would indicate an improvement in the motor-based estimate of the subject's cognitive processing speed. The 3 months off-treatment period was designed to study whether the impact of treatment persists or goes back to baseline. The number of participants that showed a decrease in the WMI score after 3 months off treatment as compared to 6 months on treatment was calculated.
Time Frame: Change after 3 months off-treatment
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 13
Participants | 7

7. Secondary Outcome: EEG Changes: Generalized Spike Wave Activity and Burst
Description: The number of generalized spike wave (GSW) activity and bursts were extracted from the patient EEGs. GSW and bursts per hour was calculated. A decrease in the spike wave and burst indicated an improvement. The number of patients that displayed a decrease in GSW and burst per hour after 6 months of treatment in noted here.
Time Frame: Change post 6 months of treatment
Population: Out of 45 enrolled, 29 patients completed the 6 month treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 29
Participants
  GSW/hr | 10
  Bursts/hr | 7

8. Secondary Outcome: EEG Changes: Generalized Spike Wave Activity and Burst
Description: The number of generalized spike wave (GSW) activity and bursts were extracted from the patient EEGs. GSW and bursts per hour was calculated. A decrease in the spike wave and burst indicated an improvement. The off-treatment period of 3 months was implemented to study whether the impact of treatment persists or goes back to baseline. The number of patients that displayed an increase in GSW and burst per hour (towards baseline) after 3 months off treatment as compared to 6 months on treatment is noted here.
Time Frame: Change after 3 months off-treatment
Population: Out of 29 patients who completed the treatment period, 28 returned for the 3 month off-treatment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 28
Participants
  GSW/hr | 13
  Bursts/hr | 11

9. Secondary Outcome: Brief Ataxia Rating Scale
Description: Ataxia is scored as per the Brief ataxia rating scale (BARS) - a modified form of the International Cooperative Ataxia Rating Scale (ICARS). The possible range for the scores is from 0 (normal, no ataxia) to 30 (severe ataxia). A decrease in the BARS score indicates an improvement in the ataxia symptoms. The number of participants that showed a decrease in BARS score after 6 months of intervention is reported here.
Time Frame: Change post 6 months of treatment
Population: Although 29 patients completed the study, some patients were unable to perform the test due to physical impairment and inability to comprehend the task. Here, the number of participants analyzed reflects the total number of patients that were present at the test and were able to complete it.
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 27
Participants | 13

10. Secondary Outcome: Brief Ataxia Rating Scale
Description: Ataxia is scored as per the Brief ataxia rating scale (BARS) - a modified form of the International Cooperative Ataxia Rating Scale (ICARS). The possible range for the scores is from 0 (normal, no ataxia) to 30 (severe ataxia). A decrease in the BARS score indicates an improvement in the ataxia symptoms. The off-treatment period of 3 months was implemented to study whether the impact of treatment persists or goes back to baseline. The number of participants that showed a subsequent increase in BARS score (towards baseline) after the of 3 months of no treatment as compared to 6 months on treatment are recorded here.
Time Frame: Change after 3 months off treatment
Population: Although 28 patients completed the off-treatment phase of study, some patients were unable to perform the test due to physical impairment and inability to comprehend the task. Here, the number of participants analyzed reflects the total number of patients that were present at the test and were able to comprehend it.
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 26
Participants | 11

11. Secondary Outcome: Clinical Global Impression Severity Scale
Description: The Clinical global impression - Severity (CGI-S) scale is used to evaluate the illness severity where the scores range from 1 (very much improved) through to 7 (very much worse). A decrease in the CGI-S score indicates a decrease in illness severity. The number of participants that showed a decrease in CGI-S score after 6 months of intervention as compared to baseline is reported here.
Time Frame: Change post 6 months of treatment
Population: Out of the 45 patients enrolled, 29 completed the 6 month treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 29
Participants | 10

12. Secondary Outcome: Clinical Global Impression Severity Scale
Description: The Clinical global impression - Severity (CGI-S) scale is used to evaluate the illness severity where the scores range from 1 (very much improved) through to 7 (very much worse). A decrease in the CGI-S score indicates a decrease in illness severity. The off-treatment period of 3 months was designed to study whether the impact of treatment persists or goes back to baseline. The number of participants that showed an increase in CGI-S score (towards baseline) after 3 months off treatment as compared to 6 months on treatment is reported
Time Frame: Change after 3 months off-treatment
Population: Out of the 29 patients that completed the treatment phase, 28 completed the following 3 month off-treatment phase. The assessment was incomplete for one patient due to inability to report symptoms.
Measure: Count of Participants; unit: Participants
Arm/Group | Triheptanoin
Number analyzed (Participants) | 27
Participants | 9

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Triheptanoin
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 41/45
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Triheptanoin (N=45)
Mild nausea (Gastrointestinal disorders) | 9
Mild vomiting (Gastrointestinal disorders) | 22
Diarrhea (Gastrointestinal disorders) | 29
Upset stomach (Gastrointestinal disorders) | 10
Stomach pain or cramping (General disorders) | 10
Acid reflux (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Seizure (Nervous system disorders) | 7
Hypoglycemia (General disorders) | 2
Loss of appetite (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT03181399/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT03181399/ICF_001.pdf